CLINICAL TRIAL: NCT01127269
Title: Practical Implementation of ADA/EASD Consensus Algorithm in Patients With Type 2 Diabetes: Timely Insulin Initiation and Titration
Brief Title: Safety and Effectiveness Study of Insulin Glargine (LANTUS) Initiation and Titration in Patients With Type 2 Diabetes
Acronym: AFICIONADO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04980; U1111-1116-9268 (Other: UTN)
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Glargine (Experimental): Patients will receive insulin glargine titrated based on standard of care as recommended by the ADA/EASD Consensus Algorithm. Step 1: insulin glargine initiation regimen for insulin naive patients/ Switch to insulin glargine for patient already treated with basal insulin.
  Step 2: the insulin dosage of patients will be titrated according to the ADA/EASD Consensus Algorithm.
  Interventions: Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous injection Dose regimen: 100 Units/mL solution for injection in a pre-filled SoloStar pen (3 ml)

SUMMARY:
Primary Objective:

Percentage of patients achieving Glycosylated Hemoglobin (HbA1c) < 7% with no severe or nocturnal hypoglycemic episodes at 6 months

Secondary Objectives:

* Glycosylated Hemoglobin (HbA1c) change from baseline to 6 months
* Insulin glargine dose at 3 and 6 months
* Hypoglycemic episodes (all types)

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of type 2 diabetes for more than 6 months
* Patients treated with Oral AntiDiabetics (OADs monotherapy or combination) with an HbA1c >7% and <10% and/or treated with NPH insulin with HbA1c >7% and <10% or treated with NPH insulin who have experienced severe and/or nocturnal hypoglycemia in the last 6 months.
* Ability to perform SMBS and insulin self-titration under the physicians guidance.
* Body Mass Index (BMI) >21 kg/ m2.
* Signature of informed consent.

Exclusion criteria:

* Hospitalized patients.
* Pregnant women or with the intention of becoming pregnant.
* Unexplained weight loss of more than 10% in the last 6 months.
* Women with child bearing potential not using effective contraceptive methods.
* Women in breast feeding period.
* Patients on chronic treatment with systemic corticosteroids or protease inhibitors.
* History of drug or alcohol abuse.
* Diabetic retinopathy with surgical treatment in 3 months previous to study entry or patients that could require surgical treatment in the following 6 months to study entry.
* Major systemic disease clinically important that would interfere with implementation or interpretation of the study, at the discretion of the investigator.
* Renal failure known as creatinine > 1.4 mg/dl in women and > 1.5 mg/dl in men.
* Known hypersensitivity to glargine or any of its excipients.
* Patients with history of hospitalization due to cardiovascular event, cardiovascular procedure in the past 6 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Glycosylated Haemoglobin (HbA1c) <7% with no severe documented nocturnal hypoglycemia episode. | From week 0 (baseline) to week 24 (end of study)

SECONDARY OUTCOMES:
Glycosylated Haemoglobin (HbA1c) | From week 0 (baseline) to week 24 (end of study)
Dose and timing of insulin glargine | From week 0 (baseline) to week 24 (end of study)
Hypoglycemic episodes | From week 0 (baseline) to week 24 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- Argentina (23):
  - Investigational Site Number 10, C.a.b.a.
  - Investigational Site Number 14, C.a.b.a.
  - Investigational Site Number 01, C.a.b.a.
  - Investigational Site Number 11, C.a.b.a.
  - Investigational Site Number 12, C.a.b.a.
  - Investigational Site Number 17, C.a.b.a.
  - Investigational Site Number 9, C.a.b.a.
  - Investigational Site Number 03, Caba
  - Investigational Site Number 06, Caba
  - Investigational Site Number 15, Caba
  - Investigational Site Number 16, Caba
  - Investigational Site Number 18, Caba
  - Investigational Site Number 26, Capital Federal
  - Investigational Site Number 22, Mar del Plata
  - Investigational Site Number 13, Mar del Plata
  - Investigational Site Number 02, Mar del Plata
  - Investigational Site Number 021, Moreno -Pcia. de Bs. As.-
  - Investigational Site Number 07, Morón
  - Investigational Site Number 04, Paraná
  - Investigational Site Number 8, Salta
  - Investigational Site Number 05, Sarandí
  - Investigational Site Number 20, Tandil
  - Investigational Site Number 25, Zárate